CLINICAL TRIAL: NCT05091268
Title: Effect of Physical Activity and Pain Education on Endometriosis-associated Pain A Randomizes Controlled Trial With a Multimodal Interdisciplinary Group Approach
Brief Title: Effect of Physical Activity and Pain Education on Endometriosis-associated Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Fysiofondet (Other); Kristiania University College (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Merete Kolberg Tennfjord, Phd, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/28494(REK)
Record Dates: First submitted 2021-09-23; First posted 2021-10-25 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Endometriosis
Keywords: endometriosis; women's health; pelvic floor; physical activity; pain education; quality of life
MeSH Terms: conditions — Endometriosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): All participants will attend a four-hour pain education session including gynecologist, psychologist, sexologist, and physiotherapist at Akershus University Hospital.
  The education will be held twice, with half of the participants at the time. The training group will then attend a 60 minutes weekly group training session led by a physiotherapist with specialist training in women's health, over a period of four months. In addition, participants will perform a progressive home exercise program performed daily over the same period. The focus will be general strength training using own body weight and cardiovascular fitness (walking, low-impact aerobic exercise), stretching, and relaxation.
  Interventions: Behavioral: Exercise
- Pain education group (No Intervention): No further follow-up

INTERVENTIONS:
Behavioral: Exercise — All participants will attend a four-hour pain education session including gynecologist, psychologist, sexologist, and physiotherapist at Akershus University Hospital.
  The education will be held twice, with half of the participants at the time. The training group will then attend a 60 minutes weekly group training session led by a physiotherapist with specialist training in women's health over a period of four months. In addition, participants will perform a progressive home exercise program performed daily over the same period. The focus will be general strength training using own body weight and cardiovascular fitness (walking, low-impact aerobic exercise), stretching, and relaxation
  Arms: Exercise group

SUMMARY:
Endometriosis is a benign gynecological condition where the uterine endometrium is located outside the uterus. The condition affects up to 10% of women of fertile age and up to 70% of women with endometriosis have symptoms with severe pain during menstruation (dysmenorrhea), pain during intercourse (dyspareunia), and/or chronic pelvic pain. Current treatments are dictated by the primary symptom: pain and are limited to surgery and hormonal treatments with often short-lived effects. Advances in the understanding of the condition have expanded to focus on less invasive and non-pharmacological treatments. Systematic reviews and meta-analyses of observational studies have focused on the protective role of physical activity and exercise on the risk of developing endometriosis. The results from these studies have been inconclusive. However, the efficacy of physical activity and exercise on pain among women with endometriosis has not been tested in high-quality randomized controlled trials (RCT).

DETAILED DESCRIPTION:
Due to the complexity of the disease, international clinical guidelines recommend that the treatment of endometriosis-associated pain should come from a multimodal and multidisciplinary perspective. Numerous non-pharmacological treatments have been proposed to alleviate endometriosis-associated pain, such as physical activity. Physical activity was introduced as a factor in the treatment of endometriosis-associated pain over three decades ago, with the possible beneficial effect that physical activity stimulates anti-inflammatory properties that will impede the development of endometriosis and lower the pain. A recent systematic review and meta-analysis found one randomized controlled study that showed no effect of physical activity on endometriosis-associated pain. They concluded that the methodological quality of this study was low, and the need for future randomized controlled studies was warranted. We, therefore, aimed to study the effect of pain education and group-based physical activity versus pain education alone on women with endometriosis-associated pain.

ELIGIBILITY:
Inclusion Criteria:

* Women of age 18-45 with signs of endometriosis on ultrasound and/or MRI and/or confirmed by laparoscopy with histology at Akershus University Hospital and Oslo University Hospital. Women may also be recruited through social media but must present with diagnosis of endometriosis.
* genital-pelvic pain ≥4/10 as measured on a numeric rating scale.
* able to understand and speak Norwegian language
* able to meet at Akershus University Hospital for participation in the study
* giving signed consent to participate.

Exclusion Criteria:

* Intra-abdominal or vaginal surgery in the last six months
* Patients who have received Botox over the past four months
* Severe pathology (malignancy),cardiovascular conditions and immune system diseases diagnosed by specialist; pregnancy, as well as childbirth the last 12 months and breastfeeding; severe psychiatric disorders that demands or has demanded admission to the hospital; personality disorder diagnosed by specialist and recently started or recently adjusted ongoing hormonal therapy.
* Participants should not have any disease or injury that could prevent them from participating in the intervention.
* Participants will be encouraged not to start with any new treatment (non-pharmacological or pharmacological) during the four-month intervention period.
* Participants who have recently undergone surgery and received Botox injections into the pelvic area can be referred but must wait 4-6 months before being included in the study. Women with planned surgery or Botox in the study period will be excluded.
* Participants recently started or adjusting ongoing hormonal therapy must wait 3-6 months to be included in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study is on endometriosis which only affect women in fertile age
Enrollment: 83 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Endometriosis associated pain | Measured at baseline and after 4 months and 12 months
  Electronically patient-reported pelvic and genital pain will include a pain body map and pain intensity scale (NRS). We will ask for average pain, worst pain, and conditional pain over the course of one month.

SECONDARY OUTCOMES:
Level of physical activity | Measured at baseline and after 4 months and 12 months
  Electronically patient-reported physical activity level will be measured using the International physical activity questionnaire-short form (IPAQ-SF). We will analyse MET values and categories of activity in addition to walking
Pelvic floor muscle maximal contraction and resting tension | Measured at baseline and after 4 months
  Pelvic floor muscle maximal contraction and muscular endurance will be measured with manometer using a vaginal balloon catheter Camtech Sandvika Norge AS (cmH2O) will be assessed. This method has demonstrated good validity and reliability, by our research group.
  Resting tension and the ability to contract using surface electromyography (EMG) will be used with a vaginal probe (Quintet). We will also perform vaginal palpation to assess pain/tenderness and tone. (All women will be instructed on how to correctly perform a pelvic floor muscle contraction prior to assessment).
Sexual function and sexual pain | Measured at baseline and after 4 months and 12 months
  Electronically patient-reported assessment using the Female Sexual Function Index (FSFI). We will also use questions adapted from Sahlgrenska University Hospital related to sexual pain. Higher scores indicates more problems. range 0-36
Depression and anxiety | Measured at baseline and after 4 months and 12 months
  Electronically patient-reported assessment using Hopkins Symptom Check List (SCL-5). Hopkins Symptom Checklist (SCL-5) was used to evaluate psychological distress, a higher score (up to 20) indicating greater psychological distress. range 0-20
Pain with urination | Measured at baseline and after 4 months and 12 months
  Electronically patient-reported assessment of pain prior to, during or after urination (developed by urologists at Akershus University Hospital). Categories of answers. Alternatives will be yes/no. questions will also cover if the symptom increases during menstruation with alternatives yes, no, sometimes, always
Bowel function | Measured at baseline and after 4 months and 12 months
  Electronically patient-reported assessment of bowel function including pain and constipation using the Knowles-Eccersley-Scott-Symptom (KESS). Higher scores indicating more problems. range 0-39
Health economy and related quality of life | Measured at baseline and after 4 months and 12 months
  Electronically patient-reported assessment using health-related quality of life questionnaire (EQ5D). Higher scores indicating better health. Questions also include questions on health care utilisation with categories over the last 4 weeks. Three questions on quality of life will also be included measured on a scale (0-10).
Fear of movement | Measured at baseline and after 4 months and 12 months
  Tampa scale measuring fair of movement. Fair avoidance with Tampa Scale for Kinesiophobia (TSK-13), which score ranges from 0 - 52, 4 subcategories, "subclinical" (score 13-22), "mild" (score 23-32) "moderate" (score 33-42) and "severe" (score 43-52).
Pain with defecation | Measured at baseline and after 4 months and 12 months
  Electronically patient-reported assessment of pain prior to, during or after defecation (developed by urologists at Akershus University Hospital). Categories of answers. Alternatives will be yes/no. questions will also cover if the symptom increases during menstruation with alternatives yes, no, sometimes, always
General pain | Measured at baseline and after 4 months and 12 months
  General pain will be assessed with a body map in addition to self-developed questions. Alternatives will be yes/no. questions will also cover if the symptom increases during menstruation with alternatives yes, no, sometimes, always

OTHER OUTCOMES:
Body mass index | Measured at baseline
  Weight and height will be combined to report BMI in kg/m^2. Weight will be measures wearing underwear and height will be measured against a wall wearing no shoes or heavy clothing.
Satisfaction and experience with physical activity and pain management | Measured after 4 months
  A qualitative interview with open ended questions to participants in both the intervention and control group that include satisfaction with participating and experience with physical exercise and pain management.
Satisfaction and experience with physical activity and pain management | Measured after 4 months and 12 months
  Self-defined questions on satisfaction with participation in the project

CONTACTS AND LOCATIONS:
Overall Officials: Merete Kolberg Tennfjord, Phd, Study Director — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lillestrøm, Nordbyhagen, Norway

IPD SHARING:
Plan to Share IPD: Yes
Within reasonable request, anonymised data could be shared with other researchers. Data from training diaries and transcripts from qualitative interviews will not be shared.
Supporting Information: Study Protocol
Time Frame: The data will be available from 2024 until 2031
Access Criteria: Researchers in the field of endometriosis

REFERENCES:
- [Derived] Gabrielsen R, Tellum T, Bo K, Engh ME, Frawley H, Nedregard Tveito S, Tennfjord MK. Supervised exercise and pelvic floor muscle training eases current pelvic and genital pain but not worst pelvic and genital pain in women with endometriosis: a randomised trial. J Physiother. 2025 Oct;71(4):246-253. doi: 10.1016/j.jphys.2025.09.012. Epub 2025 Sep 25. PMID 41006088
- [Derived] Kvale C, Tokovska M, Tennfjord MK. Women with endometriosis: Experiences with pain management and views on optimal healthcare through the concept of health literacy. Womens Health (Lond). 2025 Jan-Dec;21:17455057251347085. doi: 10.1177/17455057251347085. Epub 2025 Jul 21. PMID 40686285
- [Derived] Tennfjord MK, Gabrielsen R, Bo K, Engh ME, Molin M. Can general exercise training and pelvic floor muscle training be used as an empowering tool among women with endometriosis? Experiences among women with endometriosis participating in the intervention group of a randomized controlled trial. BMC Womens Health. 2024 Sep 12;24(1):505. doi: 10.1186/s12905-024-03356-w. PMID 39261815